CLINICAL TRIAL: NCT04290533
Title: HD-tDCS Over the dACC in High Trait Impulsivity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Monash University (Other)
Collaborators: Erasmus University Rotterdam (Other); ZonMw: The Netherlands Organisation for Health Research and Development (Other)
Responsible Party: Principal Investigator, Rebecca Segrave, Senior Research Fellow, Monash University
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Device Feasibility
Other Study IDs: 17612
Record Dates: First submitted 2020-02-18; First posted 2020-03-02 (Actual); Last update posted 2021-05-17 (Actual); Status verified 2021-05

CONDITIONS: Impulsive Behavior
Keywords: Impulsivity; HD-tDCS; dACC; ERN; Go/NoGo; MSIT
MeSH Terms: conditions — Impulsive Behavior

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active HD-tDCS (Experimental)
  Interventions: Device: Active High Definition transcranial Direct Current Stimulation (HD-tDCS)
- Sham HD-tDCS (Sham Comparator)
  Interventions: Device: Sham High Definition transcranial Direct Current Stimulation (HD-tDCS)

INTERVENTIONS:
Device: Active High Definition transcranial Direct Current Stimulation (HD-tDCS) — TDCS is a non-invasive neuromodulation technique that modulates membrane potentials by means of small electrical currents. Electrical currents induced by tDCS electrodes produce an electrical field that modulates the excitability of brain areas. In the present HD-tDCS montage, one anodal electrode and four return electrodes are applied. Hereby, the anodal electrode modulates the excitability of the targeted area, whereas the other 4 electrodes return electrical currents that flow away from that area. Direct currents will be transmitted through 5 circular PiStim electrodes of 3.14cm2 (Neuroelectrics, Barcelona, Spain; current density=0.32 mA/cm2) with a current intensity of 1.5 mA. The HD-tDCS session will last for 20 minutes in total, with a 60 sec ramp at the beginning and end of the session. The electrodes will be filled with conductive gel and plugged into an EEG cap, with the anode placed over Fz and the four return electrodes over Fp1, Fp2, F7, and F8 (10-20 system).
  Arms: Active HD-tDCS
Device: Sham High Definition transcranial Direct Current Stimulation (HD-tDCS) — For the sham-condition, the placement of the electrodes was identical to active HD-tDCS stimulation with the anode placed over Fz and the four return electrodes over Fp1, Fp2, F7, and F8 (10-20 system). The direct current, also transmitted through 5 circular PiStim electrodes of 3.14cm2 (Neuroelectrics, Barcelona, Spain; current density=0.32 mA/cm2), was increased in a ramp-like fashion over 60 seconds until it reached 1.5 mA. Directly after ramp-up, the current intensity was gradually switched off over 60 seconds, followed by 20 minutes without active stimulation. Sham procedures for tDCS mimic the transient skin sensation at the beginning of active HD-tDCS, without producing any conditioning effects on the brain. Consequently, participants are reliably blinded for sham tDCS.
  Arms: Sham HD-tDCS

SUMMARY:
Psychological disorders characterized by impulsivity often show alterations in dorsal anterior cingulate cortex (dACC) activity. Recent research has therefore focused on non-invasive neurostimulation therapies for the modulation of functional activity in the dACC. To date there has only been one proof-of-concept study providing evidence for modulating dACC activity with non-invasive electrical neurostimulation (e.g. transcranial electrical stimulation). Since transcranial Direct Current Stimulation (tDCS) is relatively safe, tolerable, and mobile as compared to other neurostimulation techniques, it is worthwhile looking further into the effects of tDCS on functional dACC activity. The aim of the present research is to explore whether HD-tDCS can induce changes in the dACC in individuals with high trait impulsivity (N=20) in a double-blind cross-over study. Functional changes in dACC activity will be measured by the error related negativity (ERN), which is an event related potential generated by the dACC. The ERN is less pronounced in people that score high on impulsivity. It is therefore expect enhanced ERN amplitudes after HD-tDCS over the dACC. In addition, performance on the multisource interference task will be used as measure of dACC activity. It is hypothesize that increased dACC activity will be related to decreased impulsivity in high impulsive individuals as shown by improved inhibitory control on the Go/NoGo task. The results of the study may have implications for patient populations that are characterized by impulsivity.

ELIGIBILITY:
Inclusion Criteria:

* Right-handed
* Score > 46 on SUPPS-P

Exclusion Criteria:

* Score low on trait impulsivity as determined by a score of < 47 on the SUPPS-P short form
* History of DSM-5 defined neurological illness, mental illness or traumatic brain injury,
* Currently taking any psychoactive medications,
* Have metal anywhere in the head, except the mouth. This includes metallic objects such as screws, plates and clips from surgical procedures.
* Currently pregnant or lactating,
* Being left-handed

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 23 (Actual)
Dates: Start 2019-03-04 (Actual); Primary Completion 2019-12-15 (Actual); Study Completion 2020-01-15 (Actual)

PRIMARY OUTCOMES:
Change in error related negativity (ERN) measured by electroencephalography (EEG) after active and sham HD-tDCS | Baseline, directly after (active vs. sham) HD-tDCS, and 30 min after (active vs. sham) HD-tDCS.
  To measure changes in electrophysiological measures of error processing after active vs. sham HD-tDCS
Change in NoGo N2 measured by electroencephalography (EEG) | Baseline, directly after (active vs. sham) HD-tDCS, and 30 min after (active vs. sham) HD-tDCS.
  To measure changes in electrophysiological measures of early inhibitory control processes after active vs. sham HD-tDCS
Change in NoGo P3 measured by electroencephalography (EEG) after active and sham HD-tDCS | Baseline, directly after (active vs. sham) HD-tDCS, and 30 min after (active vs. sham) HD-tDCS.
  To measure changes in electrophysiological measures of motor inhibitory control processes after active vs. sham HD-tDCS

SECONDARY OUTCOMES:
Change in percentage of correct nogo trials on Go/NoGo task after active vs. sham HD-tDCS | Baseline, directly after (active vs. sham) HD-tDCS, and 30 min after (active vs. sham) HD-tDCS.
  To measure the effect of active vs. sham HD-tDCS on accuracy on trials for which responses have to be inhibited. Represents a measure of change in inhibitory control.
Change in reaction times on Go trials during Go/NoGo task after active vs. sham HD-tDCS | Baseline, directly after (active vs. sham) HD-tDCS, and 30 min after (active vs. sham) HD-tDCS.
  To measure changes in speed of motor responses during Go/NoGo task differences after active vs. sham HD-tDCS
Change in reaction times post incorrect trials during Go/NoGo task after active vs. sham HD-tDCS | Baseline, directly after (active vs. sham) HD-tDCS, and 30 min after (active vs. sham) HD-tDCS.
  To measure the effect of active vs. sham HD-tDCS on post-error slowing as behavioural measure of error processing.
Change in interference effect on multisource interference task (MSIT) after active vs. sham HD-tDCS | Baseline, directly after (active vs. sham) HD-tDCS, and 30 min after (active vs. sham) HD-tDCS.
  The interference effect is calculated by subtracting the mean reaction time for congruent trials from the mean reaction time for incongruent trials. A larger interference effect reflects worse performance and is suggested to reflect decreased dACC activity.

OTHER OUTCOMES:
Trait impulsivity as measured by the The Short Version of the Urgency, Premeditation, Perseverance, Sensation Seeking and Positive Urgency Impulsive behaviour scale (SUPPS-P) | Baseline
  The SUPPS-P is a widely used robust validated 20-item scale that measures five dimensions of impulsive behavior: negative urgency, premeditation, perseverance, sensation seeking and positive urgency. Participants are asked to indicate how strongly or disagree they agree scale (1 = agree strongly to 4 = disagree strongly) with statements that relate to impulsive tendencies, such as "When I feel bad, I will often do things I later regret in order to make myself feel better now" and "I tend to lose control when I am in a great mood". Higher scores indicate more impulsiveness. For the current study, we used a cut-off score of 47 for high trait impulsivity. This score was determined following analysis of a large database (n = 485) of mental health questionnaires completed by a community sample as part of an ongoing Monash University BrainPark study.
Obsessional Behaviour Questionnaire-44 (OBQ-44) | Baseline
  The OBQ-44 is a validated 44-item questionnaire, that measures the degree of obsessional beliefs. Participants are asked to indicate how strongly or disagree they agree scale (1 = disagree very much to 7 = agree very much) with statements about responsibility/threat estimation (e.g. "harmful events will happen unless I am careful"), perfectionism/certainty (e.g. "I must be certain of my decisions"), and importance/control of thoughts (e.g. "having nasty thoughts means I am a terrible person"). A higher score means participants experience stronger obsessional beliefs.
Intolerance of Uncertainty Scale (IUS-12) | Baseline
  IUS-12 is a short version of the original 27-item Intolerance of Uncertainty Scale that measures responses to uncertainty, ambiguous situations, and the future. The 12 items are rated on a 5-point Likert scale ranging from 1 (not at all characteristic of me) to 5 (entirely characteristic of me). A higher score indicates more intolerance of uncertainty.
Demographic information | Baseline
  Age, Gender, years of education

CONTACTS AND LOCATIONS:
Locations (1):
- Monash University, BrainPark, Melbourne, Victoria, Australia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Verveer I, Hill AT, Franken IHA, Yucel M, van Dongen JDM, Segrave R. Modulation of control: Can HD-tDCS targeting the dACC reduce impulsivity? Brain Res. 2021 Apr 1;1756:147282. doi: 10.1016/j.brainres.2021.147282. Epub 2021 Jan 28. PMID 33515536